CLINICAL TRIAL: NCT03183414
Title: Right Ventricular Dysfunction in Cardiac Surgery
Brief Title: Right Ventricular Dysfunction in Cardiac Surgery Patients
Status: Completed | Type: Observational
Sponsor: Frisius Medisch Centrum (Other)
Responsible Party: Principal Investigator, Matty Koopmans, MSc, Frisius Medisch Centrum
Other Study IDs: nWMO 220
Record Dates: First submitted 2017-06-08; First posted 2017-06-12 (Actual); Last update posted 2019-11-26 (Actual); Status verified 2019-11

CONDITIONS: Right Ventricular Dysfunction
Keywords: cardiac surgery; transoesophageal echocardiography
MeSH Terms: conditions — Ventricular Dysfunction, Right

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- cardiac surgery patients: cardiac surgery patients with a significant peroperative aortic valve stenosis (gradient>40mmHg and/or aortic valve area <1cm2). During cardiac surgery measurements of right ventricular dysfunction were taken by echocardiography
  Interventions: Other: echocardiographic measurements

INTERVENTIONS:
Other: echocardiographic measurements — echocardiographic parameters of the RV, measured with TEE and the right ventricular ejection fraction (thermodilution)

SUMMARY:
To establish the correlation between echocardiographic parameters of the RV, measured with TEE and the right ventricular ejection fraction (thermodilution). To identify a time in the perioperative process when RV dysfunction occurs.

DETAILED DESCRIPTION:
Measurements with echocardiography were done during cardiac surgery to observe the right ventricular dysfunction in the perioperative process

ELIGIBILITY:
Inclusion Criteria:

* cardiac surgery patients
* elective, isolated aortic valve replacement or coronary artery bypass grafting in combination with aortic valve replacement

Exclusion Criteria:

* age < 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 15 cardiac surgery patients (elective, isolated aortic valve replacement or coronary artery bypass grafting in combination with aortic valve replacement) with a significant preoperative aortic valve stenosis (gradient>40mmHg and/or aortic valve area <1cm2)
Sampling Method: Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2017-09-06 (Actual); Primary Completion 2018-06-20 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
The correlation between echocardiographic parameters of the RV, measured with TEE and the RVEF measured with the pulmonary artery catheter | during cardiac surgery
  The correlation between echocardiographic parameters of the RV, measured with TEE and the RVEF measured with the pulmonary artery catheter.

CONTACTS AND LOCATIONS:
Overall Officials: Christiaan Boerma, MD, Principal Investigator — MCL
Locations (1):
- Medical Centre Leeuwarden, Leeuwarden, Netherlands

IPD SHARING:
Plan to Share IPD: No
not available, patient data is anonym